CLINICAL TRIAL: NCT00566761
Title: Combined Treatment of Intravitreous Bevacizumab and Triamcinolone for the Treatment or Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Treatment of Bevacizumab and Triamcinolone in Treatment or Macular Edema Secondary to CRVO
Acronym: MECROV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Carmen Cecilia Gonzalez Mijares, Asociación para Evitar la Ceguera en Mexico IAP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MECRVO
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion
Keywords: Macular edema; central retinal vein occlusion; bevacizumab; triamcinolone
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Bevacizumab; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab and triamcinolone — three applications monthly administrated of bevacizumab 2.5mg for group 1 and bevacizumab 2.5 mg + triamcinolone 4mg first dose followed by two of bevacizumab alone for the group 2

SUMMARY:
Treatment of macular edema secondary to central retinal vein occlusion is more effective with combined therapy of bevacizumab and triamcinolone than bevacizumab alone.

DETAILED DESCRIPTION:
Comparison of two groups with different treatment with registrations of outcome in BCVA and complications

ELIGIBILITY:
Inclusion Criteria:

* Macular edema secondary to central retinal vein occlusion
* BCVA worse than 20/40
* Central macular >250 mc with OCT

Exclusion Criteria:

* Diabetic retinopathy or other retinopathy
* Media opacity that does not allow following
* steroid responder
* diagnosed glaucoma or IOP > 21 mmHg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Changes in Best corrected visual acuity and macular edema measured with OCT | Follow up to 3 , 6 and 12 months

SECONDARY OUTCOMES:
Report treatment complications | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gonzalez-Mijares, Physician, Principal Investigator — Asociación para Evitar la Ceguera en México; Hugo Quiroz-Mercado, Retinologyst, Study Director — Asociación para Evitar la Ceguera en México; Juan Manuel Jimenez Sierra, Retinologyst, Study Chair — Asociación para Evitar la Ceguera en México; MA Martinez-Castellanos, Physician, Study Chair — Asociación para Evitar la Ceguera en México; Octavio Burgos Vejar, Physician, Study Chair — Asociación para Evitar la Ceguera en México; Raul Velez-Montoya, Physician, Study Chair — Asociación para Evitar la Ceguera en México; Ma de Lourdes Lopez Ramos, Physician, Study Chair — Asociación para Evitar la Ceguera en México; Omar Honerlager, preresident, Study Chair — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion Para Evitar la Ceguera en Mexico, Mexico City, Coyoacan, Mexico